CLINICAL TRIAL: NCT05268211
Title: Diagnostic Performance of Two Tools for Early Prediction of Acute Kidney Injury After Open-heart Surgery
Brief Title: Diagnostic Performance of Two Tools
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Medhat Mahfouz Eshak, Assitant Lectruer, Assiut University
Other Study IDs: IRB 5891
Record Dates: First submitted 2022-02-15; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: urinary oxygen partial pressure — measuring urinary oxygen partial pressure and measuring US Doppler renal resistive index

SUMMARY:
Developing new tools for early detection of AKI in open-heart surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing on-pump coronary artery bypass graft (CABG) surgery of both sexes

Exclusion Criteria:

* Age less than 18 years old and more than 80 years old. Patients with (CKD), chronic liver disease, heart failure, and not on diuretics or other medications that may affect renal function.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment of patients will be done through Assiut university Heart hospital after approval from the local ethics committee of the Faculty of Medicine, Assiut University
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | up to 48 hours
  Incidence of AKI according to AKIN criteria
Urinary oxygen partial pressure | up to 48 hours
  Urinary oxygen partial pressure measured in mmHg at induction, before rewarming and in the ICU
Renal resistive index | up to 48 hours
  Renal resistive index measured at induction and in the ICU